CLINICAL TRIAL: NCT05111054
Title: Sex Differences in Resistance Exercise-induced Muscle Damage: The Impact of Exercise Load
Brief Title: Sex Differences in Muscle Damage Following Resistance Exercise at Low or High Intensity
Acronym: EIMD-LOAD
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Time availability within PhD studentship
Sponsor: Durham University (Other)
Responsible Party: Principal Investigator, Alice Pearson, Principal Investigator, Durham University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 290580-LOAD
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Muscle Damage
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Load (Experimental): Acute resistance exercise performed at 30% 1RM
  Interventions: Other: Resistance Exercise
- High-Load (Active Comparator): Acute resistance exercise performed at 80% 1RM
  Interventions: Other: Resistance Exercise

INTERVENTIONS:
Other: Resistance Exercise — Acute leg-based resistance exercise bout (3 sets performed to volitional failure on leg extension and leg curl machines)

SUMMARY:
Purpose: To investigate the impact of exercise load on resistance exercise-induced muscle damage in untrained males and females.

Rationale: Unaccustomed resistance exercise can cause muscle damage, presenting as muscle soreness and reduced muscle function - such as loss of strength, power, and flexibility - for several days after the exercise bout. Therefore, individuals may require longer recovery periods before performing another exercise bout, and their performance may be impaired. Further, muscle soreness may reduce exercise compliance, particularly in novice individuals. Over time, this may compromise the gains in muscle mass and strength achieved through exercise training. Therefore, strategies to reduce the severity of exercise-induced muscle damage and/or to enhance post-exercise recovery processes are advantageous for exercising individuals.

One such strategy is to perform resistance exercise with lighter loads, i.e. <70% one repetition maximum (1RM). Low-load resistance training has shown to induce comparable gains in muscle mass and strength to high-load (≥70% 1RM), while being perceptively less exerting. Low-load resistance exercise may place less mechanical stress on muscle fibres and accordingly, its impact on muscle damage has been investigated. While several studies have reported less severe muscle damage, muscle soreness, and functional impairments with low-load resistance exercise compared to high-load, others have found no differences. Further, there is a lack of studies conducted solely in females or comparing between sexes. It has been suggested that males and females respond differently to muscle damage, and therefore, this research aims to provide a sex comparison in the muscle damage response to an acute bout of resistance exercise performed with low or high loads.

Therefore, 40 healthy, young (18-35 years) adults (20 males, 20 females) will be recruited to participate in this randomised controlled trial. Maximal leg strength and body composition (by dual-energy X-ray absorptiometry; DXA) will be conducted at baseline. In females, all primary outcome measures will be obtained during the late follicular phase of the menstrual cycle. Participants will then be randomised to a low-load (30% 1RM) or high-load (80% 1RM) exercise condition.

Three weeks later, participants will complete a resistance exercise session at their allocated intensity on leg extension and leg curl machines to induce muscle damage. Various measures of muscle damage (blood biomarkers, muscle soreness, flexibility, and swelling) will be obtained before, immediately after, and 24, 48, 72, and 168 h after the exercise protocol. The maximal strength test will be repeated 72 and 168 h after the exercise. Participants' habitual activity and dietary intake will be monitored and controlled throughout the study period.

Expected outcome: It is expected that the resistance exercise protocol will induce muscle damage, which will be less severe in the low-load exercise condition. It cannot be ascertained whether males and females will have the same responses to the exercise.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 - 25.0 kg/m2
* Untrained in resistance exercise
* No known chronic disease or current acute illness
* No current or recent (past 3 months) musculoskeletal injury
* No frequent use (2x per week for past month) of non-steroidal anti-inflammatory drugs, anti-oxidant supplements, polyunsaturated omega-3 fatty acids (and other substances that may alleviate muscle damage) and compliant to abstain from use during experimental period
* No recent or current engagement in massage or cryotherapy and compliant to abstain from use during experimental period
* Females will be eumenorrheic (regular menstrual cycle) >12 months
* Absence of pregnancy and breast-feeding

Exclusion Criteria:

* Underweight
* Overweight/obese
* Resistance trained
* Current or recent injury
* Pregnancy or breast-feeding
* Unwilling to provide blood samples, perform resistance exercise, or abstain from use of NSAID's and other substances (stated above)
* Unwilling to abstain from other forms of exercise during the experimental period

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Maximal Voluntary Contraction at baseline | Baseline
  One-repetition maximum (1RM) test: leg extension and leg curl machines
Change from baseline Maximal Voluntary Contraction at 72-hours post-exercise | 72-hours after the exercise bout
  One-repetition maximum (1RM) test: leg extension and leg curl machines
Change from baseline Maximal Voluntary Contraction at 168-hours post-exercise | 168-hours after the exercise bout
  One-repetition maximum (1RM) test: leg extension and leg curl machines
Creatine kinase concentration at baseline | Immediately pre-exercise
  Serum concentration of creatine kinase from venous blood sampling
Change from baseline in Creatine Kinase concentration immediately post-exercise | Immediately after the exercise bout
  Serum concentration of creatine kinase from venous blood sampling
Change from baseline in Creatine Kinase concentration at 24-hours post-exercise | 24-hours after the exercise bout
  Serum concentration of creatine kinase from venous blood sampling
Change from baseline in Creatine Kinase concentration at 48-hours post-exercise | 48-hours after the exercise bout
  Serum concentration of creatine kinase from venous blood sampling
Change from baseline in Creatine Kinase concentration at 72-hours post-exercise | 72-hours after the exercise bout
  Serum concentration of creatine kinase from venous blood sampling
Change from baseline in Creatine Kinase concentration at 168-hours post-exercise | 168-hours after the exercise bout
  Serum concentration of creatine kinase from venous blood sampling
Interleukin-6 concentration at baseline | Immediately pre-exercise
  Serum concentration of Interleukin-6 from venous blood sampling
Change from baseline in Interleukin-6 concentration immediately post-exercise | Immediately after the exercise bout
  Serum concentration of Interleukin-6 from venous blood sampling
Change from baseline in Interleukin-6 concentration at 24-hours post-exercise | 24-hours after the exercise bout
  Serum concentration of Interleukin-6 from venous blood sampling
Change from baseline in Interleukin-6 concentration at 48-hours post-exercise | 48-hours after the exercise bout
  Serum concentration of Interleukin-6 from venous blood sampling
Change from baseline in Interleukin-6 concentration at 72-hours post-exercise | 72-hours after the exercise bout
  Serum concentration of Interleukin-6 from venous blood sampling
Change from baseline in Interleukin-6 concentration at 168-hours post-exercise | 168-hours after the exercise bout
  Serum concentration of Interleukin-6 from venous blood sampling
Muscle soreness (pressure algometry) at baseline | Immediately pre-exercise
  Self-perceived rating of muscle soreness with use of pressure algometry
Change in muscle soreness (pressure algometry) immediately post-exercise | Immediately after the exercise bout
  Self-perceived rating of muscle soreness with use of pressure algometry
Change in muscle soreness (pressure algometry) at 24-hours post-exercise | 24-hours after the exercise bout
  Self-perceived rating of muscle soreness with use of pressure algometry
Change in muscle soreness (pressure algometry) at 48-hours post-exercise | 48-hours after the exercise bout
  Self-perceived rating of muscle soreness with use of pressure algometry
Change in muscle soreness (pressure algometry) at 72-hours post-exercise | 72-hours after the exercise bout
  Self-perceived rating of muscle soreness with use of pressure algometry
Change in muscle soreness (pressure algometry) at 168-hours post-exercise | 168-hours after the exercise bout
  Self-perceived rating of muscle soreness with use of pressure algometry
Muscle soreness (visual analogue scale, VAS) at baseline | Immediately pre-exercise
  Self-perceived rating of muscle soreness while performing a bodyweight squat with use of a visual analogue scale (0 - not sore at all, 10 - extremely sore)
Change in muscle soreness (visual analogue scale, VAS) immediately post-exercise | Immediately after the exercise bout
  Self-perceived rating of muscle soreness while performing a bodyweight squat with use of a visual analogue scale (0 - not sore at all, 10 - extremely sore)
Change in muscle soreness (visual analogue scale, VAS) at 24-hours post-exercise | 24-hours after the exercise bout
  Self-perceived rating of muscle soreness while performing a bodyweight squat with use of a visual analogue scale (0 - not sore at all, 10 - extremely sore)
Change in muscle soreness (visual analogue scale, VAS) at 48-hours post-exercise | 48-hours after the exercise bout
  Self-perceived rating of muscle soreness while performing a bodyweight squat with use of a visual analogue scale (0 - not sore at all, 10 - extremely sore)
Change in muscle soreness (visual analogue scale, VAS) at 72-hours post-exercise | 72-hours after the exercise bout
  Self-perceived rating of muscle soreness while performing a bodyweight squat with use of a visual analogue scale (0 - not sore at all, 10 - extremely sore)
Change in muscle soreness (visual analogue scale, VAS) at 168-hours post-exercise | 168-hours after the exercise bout
  Self-perceived rating of muscle soreness while performing a bodyweight squat with use of a visual analogue scale (0 - not sore at all, 10 - extremely sore)
Range of motion at baseline | Immediately pre-exercise
  Flexibility of the exercised limb as determined by goniometry
Change in range of motion immediately post-exercise | Immediately after the exercise bout
  Flexibility of the exercised limb as determined by goniometry
Change in range of motion at 24-hours post-exercise | 24-hours after the exercise bout
  Flexibility of the exercised limb as determined by goniometry
Change in range of motion at 48-hours post-exercise | 48-hours after the exercise bout
  Flexibility of the exercised limb as determined by goniometry
Change in range of motion at 72-hours post-exercise | 72-hours after the exercise bout
  Flexibility of the exercised limb as determined by goniometry
Change in range of motion at 168-hours post-exercise | 168-hours after the exercise bout
  Flexibility of the exercised limb as determined by goniometry
Limb circumference at baseline | Immediately pre-exercise
  Measure of leg circumference with use of standard anthropometric tape to indicate muscle swelling
Change in limb circumference immediately post-exercise | Immediately after the exercise bout
  Measure of leg circumference with use of standard anthropometric tape to indicate muscle swelling
Change in limb circumference at 24-hours post-exercise | 24-hours after the exercise bout
  Measure of leg circumference with use of standard anthropometric tape to indicate muscle swelling
Change in limb circumference at 48-hours post-exercise | 48-hours after the exercise bout
  Measure of leg circumference with use of standard anthropometric tape to indicate muscle swelling
Change in limb circumference at 72-hours post-exercise | 72-hours after the exercise bout
  Measure of leg circumference with use of standard anthropometric tape to indicate muscle swelling
Change in limb circumference at 168-hours post-exercise | 168-hours after the exercise bout
  Measure of leg circumference with use of standard anthropometric tape to indicate muscle swelling

CONTACTS AND LOCATIONS:
Overall Officials: Alice G Pearson, Principal Investigator — Durham University
Locations (1):
- Durham University, The Graham Sports Centre, Durham, County Durham, United Kingdom